CLINICAL TRIAL: NCT00653315
Title: To Compare the Relative Bioavailability of the Kali's Tramadol APAP Tablets With Ortho-McNeil's Ultracet Tablets Under Fasting Conditions.
Brief Title: Bioavailability Study of Tramadol/APAP Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: AAI Clinic (Other)
Responsible Party: Alfred Elvin// Director Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-121
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: To Determine Bioequivalence Under Fasting Conditions
Keywords: Bioequivalence, Tramadol APAP, fasting
MeSH Terms: conditions — Fasting | interventions — Ultracet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received kali product under fasting conditions
  Interventions: Drug: Tramadol APAP
- B (Active Comparator): Subjects received Ortho-Mcneil product under fasting conditions
  Interventions: Drug: Ultracet

INTERVENTIONS:
Drug: Tramadol APAP — Tablets, 37.5mg/325mg, single dose
  Other Names: Ultracet
  Arms: A
Drug: Ultracet — Tablets, 37.5mg/325mg
  Other Names: Tramadol APAP
  Arms: B

SUMMARY:
To compare the relative bioavailability of Kali and Ortho-McNeil's

DETAILED DESCRIPTION:
To compare the relative bioavailability of Kali's Tramadol/APAP 37.5mg/325mg with Ortho-McNeil's Ultracet tablets 37.5mg/325mg

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and females between 18 and 45 years of age inclusive
* Informed of the nature of the study and given written informed consent.
* Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables and weighing at least 100lbs.

Exclusion Criteria:

* Hypersensitivity to Tramadol/ Acetaminophen, opioids such as morphine and codeine, or related compounds, or a history or seizures.
* Any history of a clinical condition which might affect drug absorption, metabolism or excretion.
* Recent history (within one year) of mental illness, drug illness, drug abuse or alcoholism.
* Donation of greater than 500mL of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
* Received an investigational drug within the 4 weeks prior to study dosing.
* Currently taking any prescription medication, except oral contraceptives, within 7days prior to study dosing or over-the-counter medication within 3 days of the study dosing.
* This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the physician.
* Tobacco use(>5 cigarettes per day)in the 3 months prior to study dosing.
* If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the two treatment periods.
* Females of child bearing potential must use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed.
* Medically acceptable methods of contraception that may be used by the subject and/or her partner are:oral contraceptive, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence.
* females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2002-05; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of absorption | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Scallion, Principal Investigator — AAI Clinic